CLINICAL TRIAL: NCT03838874
Title: Double Blind Randomized Clinical Trial Comparing Time To Return of Lower Extremity Motor Function Following Spinal Anesthetic With Mepivacaine Versus Low-Dose Bupivacaine For Primary Total Hip and Knee Arthroplasty
Brief Title: Mepivacaine Versus Low-Dose Bupivacaine For Primary Total Hip and Knee Arthroplasty
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew P. Abdel, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-008635
Record Dates: First submitted 2019-02-11; First posted 2019-02-12 (Actual); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Bupivacaine; Mepivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-Dose Bupivacaine (Active Comparator): Subjects in this group will be given 10mg of Low-Dose Bupivacaine, which is within standard of care for spinal anesthesia during TKA or THA.
  Interventions: Drug: Low-Dose Bupivacaine
- Mepivacaine (Active Comparator): Subjects in this group will be given 70mg of Mepivacaine, which is within standard of care for spinal anesthesia during TKA or THA.
  Interventions: Drug: Mepivacaine

INTERVENTIONS:
Drug: Low-Dose Bupivacaine — 10 mg (2 mL of 0.5%) administered as an isobaric spinal anesthetic
  Arms: Low-Dose Bupivacaine
Drug: Mepivacaine — 70 mg (3.5 mL of 2%) administered as an isobaric spinal anesthetic
  Arms: Mepivacaine

SUMMARY:
This research is being done to see if there is a difference between two different spinal anesthetics (Mepivacaine vs. Bupivacaine) as it relates to reducing post-operative complications and the time it takes for subjects to regain mobility after surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physiological status I-III (patient must meet criteria of a status I-III in the ASA Physical Status Classification System: I=Normal Healthy Patient, II=Mild Systemic Disease, and III=Severe Systemic Disease)
* Unilateral primary TKA or THA
* 18+ years of age
* Able to provide informed consent

Exclusion Criteria:

* Chronic pain syndromes such as fibromyalgia or complex regional pain syndrome
* Chronic opioid use (>1 mos) with OME >5 mg/day OR acute opioid use (< 1 mos) with OME > 30 mg/day.
* Body mass index (BMI) > 45 kg/m2
* Severe drug allergy* to medications used in this study, including non-steroidal anti-inflammatory drugs (i.e. celecoxib and ketorolac), and local anesthetics (defined as an immune reaction resulting in shortness of breath, hives, anaphylaxis, wheezing, and fever)
* Major systemic medical comorbidities such as:

  * Pre-existing severe renal disorder defined as glomerular filtration rate (GFR) <50 units/m2 (if labs are available), currently on dialysis, or highly suspected based on history.
  * Severe hepatic disorder defined as current or past diagnosis of acute/subacute necrosis of liver, acute hepatic failure, chronic liver disease, cirrhosis (primary biliary cirrhosis), chronic hepatitis/toxic hepatitis, liver abscess, hepatic coma, hepatorenal syndrome, other disorders of liver
* Contraindication to spinal anesthesia technique (e.g., known spinal stenosis, coagulopathy, sepsis, infection at site of injection, uncooperative, refusal, anticoagulation medications not held within appropriate time frame*). *Per ASRA guidelines, Clopidogrel (Plavix) held for at least 7 days, Dabigatran (Pradexa) held for at least 5 days, Rivaroxaban (Xarelto)held for at least 3 days, Warfarin (Coumadin)held for at least 5 days or recent INR of less than 1.4, Enoxaparin (Lovenox) with doses > 1 mg/kg held for close to 24 hours.
* Known to be currently pregnant or actively breastfeeding. Patients that have a previous history of menopause, hysterectomy, or tubal ligation will not be required to perform a pregnancy test. Female patients that do not meet this criterion will be asked to submit a urine sample, and will require a negative urine sample in order to proceed with study protocol. Urine sample be collected pre-procedurally.
* Impaired cognition

Min Age: 18 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Abdel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-Dose Bupivacaine | Mepivacaine
Started | 80 | 74
Completed | 80 | 74
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Dose Bupivacaine | Mepivacaine | Total
Number analyzed (Participants) | 80 | 74 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (11.8) | 67.9 (9.2) | 67.9 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 42 | 88
  Male | 34 | 32 | 66
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 80 | 74 | 154

OUTCOME MEASURES:

1. Primary Outcome: Time to Return of Lower Extremity Motor Function
Description: Assessed by measuring time from spinal anesthetic administration to postoperative achievement of Bromage 0 function (return of spontaneous ankle, knee, and hip movement) in the non-operative extremity at 15-minute intervals.
Time Frame: Post surgery, approximately 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Low-Dose Bupivacaine | Mepivacaine
Number analyzed (Participants) | 80 | 74
minutes | 210.3 (79.54) | 184.7 (47.8)

2. Secondary Outcome: Post-Anesthesia Care Unit (PACU) Length of Stay
Description: Number of minutes subjects were admitted to PACU following the surgical procedure
Time Frame: Time of discharge, approximately 1-2 days
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Low-Dose Bupivacaine | Mepivacaine
Number analyzed (Participants) | 80 | 74
minutes | 65.2 (33.6) | 75.0 (39.3)

3. Secondary Outcome: Hospital Length of Stay
Description: Number days subjects were admitted to the hospital following the surgical procedure
Time Frame: Time of discharge, approximately 1-2 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Low-Dose Bupivacaine | Mepivacaine
Number analyzed (Participants) | 80 | 74
days | 1.5 (0.9) | 1.4 (0.8)

4. Secondary Outcome: Maximum Pain Score
Description: Measured on a scale from 1 to 10 in the first 24 hours following the surgical procedure, 1=mild pain; 10=worst pain.
Time Frame: 24 hours following the surgical procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-Dose Bupivacaine | Mepivacaine
Number analyzed (Participants) | 80 | 74
score on a scale | 6.0 (2.5) | 6.5 (2.1)

5. Secondary Outcome: Median Pain Score
Description: Measured on a scale from 1 to 10 in the first 24 hours following the surgical procedure, 1=mild pain; 10=worst pain.
Time Frame: 24 hours following the surgical procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-Dose Bupivacaine | Mepivacaine
Number analyzed (Participants) | 80 | 74
score on a scale | 3.4 (1.9) | 3.4 (1.6)

6. Secondary Outcome: Discharge Pain Score
Description: Measured on a scale from 1 to 10 at time of hospital discharge, 1=mild pain; 10=worst pain.
Time Frame: Time of discharge, approximately 1-2 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-Dose Bupivacaine | Mepivacaine
Number analyzed (Participants) | 80 | 74
score on a scale | 3.5 (2.1) | 3.5 (2.1)

7. Secondary Outcome: Orthostatic Hypotension
Description: Number of participants to experience orthostatic hypotension following the surgical procedure.
Time Frame: Time of discharge, approximately 1-2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low-Dose Bupivacaine | Mepivacaine
Number analyzed (Participants) | 80 | 74
Participants | 4 | 6

8. Secondary Outcome: Urinary Retention
Description: Number of participants to experience urinary retention follow the surgical procedure.
Time Frame: Time of discharge, approximately 1-2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low-Dose Bupivacaine | Mepivacaine
Number analyzed (Participants) | 80 | 74
Participants | 10 | 10

9. Secondary Outcome: Transient Neurologic Symptoms
Description: Number of participants to report transient neurologic symptoms
Time Frame: One week post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Low-Dose Bupivacaine | Mepivacaine
Number analyzed (Participants) | 80 | 74
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 6-9 days on all participants.
Arm/Group | Low-Dose Bupivacaine | Mepivacaine
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/74
Other Adverse Events (participants affected / at risk) | 0/80 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT03838874/Prot_SAP_000.pdf